CLINICAL TRIAL: NCT06785194
Title: Samfilcon B Custom Toric Lens Real-World Observational Study
Brief Title: Revive Toric RWE Study
Status: Not yet recruiting | Type: Observational
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: RWE-REV-P85-001
Record Dates: First submitted 2025-01-16; First posted 2025-01-21 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- REVIVE samfilcon B custom toric contact lenses: REVIVE samfilcon B custom toric contact lenses
  Interventions: Device: REVIVE samfilcon B custom toric contact lenses

INTERVENTIONS:
Device: REVIVE samfilcon B custom toric contact lenses — REVIVE samfilcon B custom toric contact lenses

SUMMARY:
This is a post-market observational clinical investigation. The objective of this observational study is to evaluate the visual performance and HCP satisfaction of REVIVE samfilcon B custom toric contact lenses.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years or older on the date the ICF is signed
2. Have the capacity to read, understand, and provide written voluntary informed consent
3. Have physiologically normal anterior segments not exhibiting clinically significant biomicroscopy findings
4. Have no active ocular disease or allergic conjunctivitis
5. Not be using any topical ocular medications
6. Be willing and able to follow instructions
7. Have signed a statement of informed consent
8. Be an experienced soft contact lens wearer (have previously used soft contact lenses)
9. Meet the indications per the Instructions for Use (IFU) and have a suitable prescription for treatment with the device

Exclusion Criteria:

1. Is participating in another research study
2. Is considered by the Investigator to not be a suitable candidate for participation
3. Is not eligible for treatment with the study lens per the IFU (contraindicated)
4. Has had previous ocular surgery
5. Is taking/using ocular, systemic, or topical medications that, in the Investigator's opinion, could potentially affect ocular physiology or lens/solution performance

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient population at study site locations
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Investigator overall satisfaction as assessed by the Investigator Survey | Assessed 14 days ± 3 days after the final dispensing/refinement visit
  (completed by the Investigator for each subject at 14 days ± 3 days after the final dispensing/refinement visit)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Site 101, Orange Park, Florida
  - Site 102, Orange Park, Florida
  - Site 103, Canton, Georgia